CLINICAL TRIAL: NCT05577728
Title: Prediction of the SEPRA Diabetes Trial in Healthcare Claims Data
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Associate Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2018P002966-DUP-SEPRA
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- New use of semaglutide injection: Exposure group
  Interventions: Drug: New use of semaglutide injection
- New initiation of "standard of care": (SGL2i, 2nd generation SU, DPP-4i and GLP-1 RA except for semaglutide inj or oral) Reference group
  Interventions: Drug: New initiation of "standard of care" (SGL2i, 2nd generation SU, DPP-4i and GLP-1 RA except for semaglutide inj or oral)

INTERVENTIONS:
Drug: New use of semaglutide injection — New use of semaglutide injection dispensing claim is used as the exposure.
  Groups: New use of semaglutide injection
Drug: New initiation of "standard of care" (SGL2i, 2nd generation SU, DPP-4i and GLP-1 RA except for semaglutide inj or oral) — New initiation of "standard of care" (SGL2i, 2nd generation SU, DPP-4i and GLP-1 RA except for semaglutide inj or oral) dispensing claim is used as the reference.
  Groups: New initiation of "standard of care"

SUMMARY:
Investigators are building an empirical evidence base for real world data through large-scale replication of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the RCT DUPLICATE initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to replicate, as closely as is possible in healthcare insurance claims data, the trial listed below/above. Although many features of the trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. Randomization is also not replicable in healthcare claims data but was proxied through a statistical balancing of measured covariates according to standard practice. Investigators assume that the RCT provides the reference standard treatment effect estimate and that failure to replicate RCT findings is indicative of the inadequacy of the healthcare claims data for replication for a range of possible reasons and does not provide information on the validity of the original RCT finding.

ELIGIBILITY:
All patients will be required to have continuous enrollment during the baseline period of 180 days before initiation of semaglutide or standard of care (SGL2i, 2nd generation SU, DPP-4i and GLP-1 RA except for semaglutide inj or oral) (cohort entry).

Eligible cohort entry dates:

Market availability of semaglutide/standard of care in the US started on December 6th, 2017:

* For Optum: December 6, 2017 - May 31, 2021 (end of data availability)

Inclusion Criteria:

* Age >= 18
* Type 2 diabetes mellitus diagnosis
* Use of metformin
* At least 2 HbA1c records within the prior 280 days
* At least 1 HbA1c record within the prior 90 days

Exclusion Criteria:

* Missing age or gender
* Use of any other anti-diabetes medications
* Any insulin use
* Pregnancy
* Multiple Endocrine Neoplasia syndrome type 2
* CKD stage 5, ESRD, dialysis, or renal transplant
* Nursing home admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes who have previously been treated with metformin.
Sampling Method: Non-Probability Sample
Enrollment: 2316 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Long-term glycemic control defined as proportion of patients who will achieve an HbA1c of less than 7.0% (53.0 mmol/mol) | At year 1
  Number of subjects

SECONDARY OUTCOMES:
Change in HbA1c | At 1 year
  Change in HbA1c from baseline at 365 days after drug initiation.
Number of hypoglycemic episodes leading to an inpatient admission or emergency room encounter. | At 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, ScM, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Kattinakere Sreedhara S, Schneeweiss S, D'Andrea E, Weberpals JG, DiCesare EC, Patorno E, Tsacogianis T, Bradley M, Concato J, Wang SV. Using real-world data to predict findings of an ongoing phase IV trial: glycemic control of semaglutide versus standard of care. BMJ Open Diabetes Res Care. 2025 Oct 29;13(5):e005180. doi: 10.1136/bmjdrc-2025-005180. PMID 41161770

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan: Study Protocol and Statistical Analysis Plan (2022-10-07): https://cdn.clinicaltrials.gov/large-docs/28/NCT05577728/Prot_SAP_000.pdf